CLINICAL TRIAL: NCT03072420
Title: Characterization of Fingertips Using MRI Images : Development of Mechanically Faithful Models Dedicated to Manipulation.
Brief Title: Characterization of Fingertips Using MRI Images (FINGERS-COMPRESSION)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0688
Record Dates: First submitted 2017-02-21; First posted 2017-03-07 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: MRI, fingers compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group no manual work or activity (Experimental): Subject with an office or student job.
  Interventions: Other: Compression of the fingertip under MRI.
- Group manual work (Sham Comparator): Subject working in a manual or predominantly manual.
  Interventions: Other: Compression of the fingertip under MRI.

INTERVENTIONS:
Other: Compression of the fingertip under MRI. — Compression of the fingertip by a static loading on the phalanx distal of the index of the subjects; Then also a shear stress in the transverse direction of the finger. The data provided by the MRI images will be geometric information such as the thickness of the skin and its possible variation as a function of the area of the finger, the total thickness of soft tissues in compression as a function of the variation in l The angle between the axis of the phalanx and the plane of contact; Mechanical type information relating to the displacements and reaction forces, to the internal deformations of the different areas of the finger.

SUMMARY:
The objectives was to obtain MRI images of the index finger of the subjects without loading and with loadings (normal and shear forces from 1 to 4N).

ELIGIBILITY:
Inclusion Criteria:

* Active voluntary healthy adult aged 18 to 65, affiliated to a social security scheme
* Stature between 170 and 179cm
* Body mass index (BMI) between 20 and 25
* No previous hand musculoskeletal disorders
* Cognitive level compatible with oral communication, adherence to instructions and understanding of gestures
* Having signed the consent to participate in the study

Exclusion Criteria:

* the subject presents a neurological or orthopedic disorder ;
* the subject presents a pathology that could disturb the task ;
* the subject has an Magnetic Resonance Imaging (MRI) contraindication (wears a pacemaker, insulin pump, prothesis, etc, has claustrophobia, …)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2015-07-24 (Actual); Study Completion 2015-07-24 (Actual)

PRIMARY OUTCOMES:
Average fingertip deflection under compression | Day 1
  The different stresses will be: compression of the fingertip by a static loading on the phalanx distal of the index of the subjects; Then also a shear stress in the transverse direction of the finger.

SECONDARY OUTCOMES:
Average fingertip dimensions | Day 1
  In order to develop realistic biomechanical models of the fingers allowing the simulation of the grip, an essential step will be the experimental mechanical characterization of the distal phalanges.

CONTACTS AND LOCATIONS:
Overall Officials: Georges BARATON, MD, Principal Investigator — IFSTTAR
Locations (1):
- IFSTTAR, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dallard J, Merlhiot X, Petitjean N, Duprey S. MRI-based experimentations of fingertip flat compression: Geometrical measurements and finite element inverse simulations to investigate material property parameters. J Biomech. 2018 Jan 23;67:166-171. doi: 10.1016/j.jbiomech.2017.11.024. Epub 2017 Nov 29. PMID 29217092